CLINICAL TRIAL: NCT00278122
Title: Evaluation of the Clinical Efficacy of Leukine® Administered in Conjunction With Paclitaxel in Patients With Advanced Melanoma
Brief Title: Paclitaxel and GM-CSF in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William W. Grosh, University of Virginia Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: 11782; UVACC-MEL-46; UVACC-HIT-028.8; UVACC-PRC-350-04
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — sargramostim; Paclitaxel

INTERVENTIONS:
Biological: sargramostim
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop tumor cells from growing. Giving paclitaxel together with GM-CSF may be effective in treating melanoma.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with GM-CSF works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the activity of paclitaxel and sargramostim (GM-CSF), in terms of objective clinical response rate (complete response [CR] and partial response [PR]), in patients with advanced unresectable melanoma.

Secondary

* Evaluate the duration of response, time to progression, and overall survival of patients treated with this regimen.
* Determine serum cytokine levels (GM-CSF, IFN-γ, aldesleukin, recombinant interleukin-4, and IL-10) in these patients.

OUTLINE: This is an open-label study.

Patients receive paclitaxel IV over 3 hours on day 1 and sargramostim (GM-CSF) subcutaneously on days 4-17. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses of therapy beyond CR for up to 12 courses.

After study treatment, patients are followed every 3-6 months for at least 3 years.

PROJECTED ACCRUAL: A total of 42 patients will accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable stage III or IV melanoma from a cutaneous, mucosal, or unknown primary site

  * Unresectable stage III disease, defined as meeting 1 of the following criteria:

    * Regional metastasis that, in the judgement of the treating physician, cannot be surgically resected with clear margins
    * Regional metastasis that can be surgically resected with clear margins only by extensive surgery that is inadvisable or unacceptable to the treating physician and/or patient
  * Staging of cutaneous and mucosal melanoma based on the revised American Joint Committee on Cancer (AJCC) staging system
* Must have measurable disease as defined by Response Evaluation Criteria in Small Tumors (RECIST) criteria
* No ocular melanoma
* Patients with brain metastases may be eligible if all of the following are true:

  * Total number of brain metastases ever is ≤ 3
  * Each brain metastasis has been completely removed by surgery or each unresected brain metastasis has been treated with stereotactic radiosurgery

    * Stereotactic radiosurgery, such as gamma knife, can be used up to 1 week before study entry
    * No evident growth of any brain metastasis since treatment
  * No brain metastasis that is > 2 cm in diameter at study entry

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin normal
* Creatinine ≤ 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No previous or concurrent autoimmune disorder requiring cytotoxic or immunosuppressive therapy
* No autoimmune disorder with visceral involvement

  * The following conditions are allowed:

    * Laboratory evidence of autoimmune disease (e.g., positive ANA titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring steroidal anti-inflammatory drugs
* HIV negative
* Hepatitis C negative
* No other serious or poorly controlled medical condition that could be exacerbated by or complicate compliance with study therapy

PRIOR CONCURRENT THERAPY:

* No more than 1 previous chemotherapy regimen for metastatic melanoma
* No previous paclitaxel
* No chemotherapy, interferon, growth factors, interleukin, or radiotherapy (excluding gamma knife therapy for brain metastases) within the past 4 weeks
* No surgical resection of metastatic lesions within the past 4 weeks
* No other investigational medication within the past 4 weeks or during study
* No nitrosoureas (e.g., carmustine or lomustine) within the past 6 weeks and during study treatment
* No other concurrent chemotherapy, interferon, other growth factors, interleukin, illegal drugs, radiotherapy, surgery, or steroid therapy
* No concurrent oral or injectable hydrocortisone (at doses > 15 mg per day) or its equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response by CT scans every 6 weeks

SECONDARY OUTCOMES:
Duration of response by CT scans every 6 weeks
Time to progression by CT scans every 6 weeks
Survival

CONTACTS AND LOCATIONS:
Overall Officials: William W. Grosh, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States